CLINICAL TRIAL: NCT01932385
Title: Phase 2 Study of Sorafenib in the Management of Liver Function Impaired Advanced Hepatocellular Carcinoma
Brief Title: Sorafenib in Liver Function Impaired Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Qingdao Central Hospital (Other)
Responsible Party: Principal Investigator, Youxin Ji, Chief, Department of Oncology, Qingdao Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QCH20130823
Record Dates: First submitted 2013-08-22; First posted 2013-08-30 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2015-10

CONDITIONS: Liver Cancer
Keywords: Sorafenib; Hepatocellular carcinoma; Best supportive care; Survival
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- sorafenib (Experimental): sorafenib 400mg, oral, twice a day until disease progression defined by RECIST.
  Interventions: Drug: Sorafenib; Other: Best Supportive Care
- Best Supportive Care (Active Comparator): treatment mainly on nutrition and symptoms control
  Interventions: Other: Best Supportive Care

INTERVENTIONS:
Drug: Sorafenib
  Other Names: Nexavar
  Arms: sorafenib
Other: Best Supportive Care

SUMMARY:
Due to the HBV and HCV infection, about 55% hepatocellular carcinoma patients happened in China. Among them, only 10% patients can be diagnosed in early stage. Sorafenib increased PFS and OS in advanced hepatocellular carcinoma patients with liver function of Child-Pugh class A patients, but the result for Child-Pugh class B patients is unclear.

ELIGIBILITY:
Inclusion Criteria:

* pathological or cytological confirmed advanced hepatocellular carcinoma
* 18 years to 80 years
* liver function Child-Pugh class B
* BCLC stage B or C
* estimated life time 2 months or longer

Exclusion Criteria:

* previous target therapy
* allergy to Sorafenib
* Uncontrolled Bleeding or diarrhea
* eligible for locoregional treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2013-08-01; Primary Completion 2016-01-30 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
progression free survival and overall survival | From date of randomization until the date of first documented progression or date of death from any cause up to 12 months

SECONDARY OUTCOMES:
response rate | every 4 weeks till progression, total up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: ketao lan, M.D., Study Director — Qingdao Health Bereau
Locations (1):
- Qingdao Central Hospital, Qingdao Cancer Hospital, Qingdao, Shandong, China